CLINICAL TRIAL: NCT02105103
Title: Accu-Chek® Insight Insulin Pump EU Study: A European Multicenter Study to Evaluate the Accu-Chek® Insight Insulin Pump in Routine Practice
Brief Title: European, Open-label, Prospective, Multinational, Multicenter Study in Adult Subjects With Type 1 or Type 2 Diabetes Previously on MDI or CSII Therapy. Subjects Home Setting is Considered Routine Practice.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RD001514
Record Dates: First submitted 2014-03-28; First posted 2014-04-07 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Type 2 Diabetes, Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1

ARMS (1):
- Accu-Chek® Insight Insulin Pump (Other)
  Interventions: Device: Accu-Chek® Insight Insulin Pump

INTERVENTIONS:
Device: Accu-Chek® Insight Insulin Pump — A new insulin pump, the Accu-Chek® Insight insulin pump, will be used by all subjects enrolled in this study. The usability of the Accu-Chek® Insight insulin pump for the intended use has already been investigated in a Human Factor study. The study subjects may encounter the following potential risks of CSII therapy while participating in the study: Possible hypoglycemia; Possible hyperglycemia which might progress to ketosis and DKA; Infusion site reactions (bleeding, bruising, discomfort, pruritus, pain, plaster reactions, inflammation, infection etc.)

SUMMARY:
Accu-Chek® Insight Insulin Pump EU Study is a Multicenter Study to evaluate the Accu-Chek® Insight Insulin Pump in routine practice. This is an open-label, prospective, multinational, multicenter study evaluating the CSII therapy with the Accu-Chek Insight Insulin pump in routine practice in adult subjects with Type 1 or type 2 diabetes. Subjects must have been on intensive insulin therapy for at least six months i.e. either on CSII or MDI. All subjects will receive training in the preparation, programming and daily use of the Accu-Chek Insight Insulin pump. In addition, subjects previously on MDI may receive more training in order to be comfortable with the use of an insulin pump. The study will be conducted in 10-12 sites in Austria, France and the United Kingdom. A total of 80-95 subjects will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years old
* Diagnosed at least for 12 months with Type 1 or 2 Diabetes requiring insulin therapy
* Intensive insulin therapy by MDI or CSII at least 6 months
* Willing to self monitor blood glucose 4 times daily

Exclusion Criteria:

* Significantly impaired awareness of hypoglycemia
* Unstable chronic disease other than diabetes
* Acute illness or inability to recognize pump signals or alarms as determined by the investigator
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
The primary objective is to evaluate the Accu-Chek Insight Insulin Pump and associated pump devices in routine practice. This will be expressed by the rate of error messages per 100 patient years (confirmed by pump uploads). | 6 months

SECONDARY OUTCOMES:
Evaluate type and frequency of adverse events (serious/non-serious) possibly related or related to study devices and/or study procedures | 6 months
Evaluate subject satisfaction based on surveys of important factors of health-related quality of life | 6 months
Evaluate change in HbA1c from screening to month 3 and 6 | 3 weeks screening plus 6 months treatment period
Evaluate utilization of pump functions (e.g. basal rate profiles, temporary basal rates, bolus types) | 6 months
Evaluate change in CGM-derived parameters from month 3 to month 6 | 6 months
Evaluate type and frequency of pump signals, i.e. reminders, errors, warnings, alarms, maintenance messages | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Petersen, Study Director — Roche Diagnostics GmbH
Locations (7):
- Austria (2):
  - Graz
  - Vienna
- United Kingdom (5):
  - Birmingham
  - Blackburn
  - Leicester
  - Middlesbrough
  - Stafford